CLINICAL TRIAL: NCT02655341
Title: Hydration Status Assessment Through Body Composition Monitoring And Renal Artery Stenosis Evaluation in Patients With Acute Myocardial Infarction Referred For Primary PCI
Brief Title: Hydration Status Assessment Through Body Composition Monitoring in Patients With Acute Myocardial Infarction
Acronym: HYD-AMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor Adrian Covic, MD, PhD, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: HYD-AMI001
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Dehydration; Acute Myocardial Infarction; Renal Artery Stenosis
Keywords: Dehydration; Primary PCI; Acute Myocardial Infarction; Bioimpedance; Renal Angiography
MeSH Terms: conditions — Dehydration; Renal Artery Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Consecutive STEMI Patients: All patients with AMI referred for primary PCI in a single centre
  Interventions: Device: Body Composition Monitoring; Procedure: Coronarography; Procedure: Primary Percutaneous Coronary Intervention; Procedure: Renal Angiography

INTERVENTIONS:
Device: Body Composition Monitoring — using Fresenius device; two measurements before and after coronary intervention;
  Other Names: BCM
Procedure: Coronarography — Preprocedural coronary arteriography is obtained after sterile preparation and draping of the patient, conscious sedation, infiltration of local anesthetic (lidocaine solution) at the femoral access site, placement of an arterial sheath in the femoral artery, and advancement of the renal guide catheter over a 0.035-in guidewire under fluoroscopic guidance. After the tip of the guide catheter is positioned at the ostium of the left coronary stem, an angiogram is obtained. After the guidewire is removed, the proximal end of the catheter is connected to a manifold, and 4-8 mL of contrast is manually injected during cineangiographic recording.
  Other Names: Coronary Artery Angiography
Procedure: Primary Percutaneous Coronary Intervention — An intravenous antithrombotic agent, usually heparin, is administered before the clinician proceeds with angioplasty.
  Other Names: Primary PCI
Procedure: Renal Angiography — After the tip of the guide catheter is positioned at the ostium of the renal artery, an angiogram is obtained. After the guidewire is removed, the proximal end of the catheter is connected to a manifold, and 4-8 mL of contrast is manually injected during cineangiographic recording. This procedure is performed in the same time with primary PCI
  Other Names: RA

SUMMARY:
Aims:

* evaluate the hydric status through bioimpedance spectroscopy in consecutive acute myocardial infarction patients referred for primary PCI;
* assessment of renal artery stenosis incidence through renal angiography in consecutive STEMI patients;
* fully characterize the complex hydration, metabolic and endothelial profile of these patients in the attempt to define the role played by dehydration in the complex dynamics of acute myocardial infarction.

DETAILED DESCRIPTION:
Gathered data:

* descriptive general demographic data;
* previous pathologies (ischemic heart disease, peripheral arterial disease, stroke, heart failure, previous percutaneous coronary interventions, coronary artery bypass grafting - CABG, known renal disease);
* cardiovascular risk factors (age, weight, height, abdominal perimeter, body mass index, smoking, sedentariness, diabetes, hypertension, dyslipidaemia);
* routine biological data;
* metabolic data (obtained from two body composition monitoring evaluations - before and 12 hours after coronary intervention) - body water, body fat tissue;
* information regarding primary PCI (less than 12 hours of ischemic symptoms);
* coronarographic details, type of used stent, periprocedural specific complications, final TIMI - thrombolysis in myocardial infarction - flow);
* echocardiography at admission (LVEF);
* renal arteries angiographic details performed in the same time with PCI (two independent operators evaluate stenosis based on a predefined scale);
* renal diameters;
* measurement of arterial stiffness through Sphigmocore pulsed-wave-velocity (24 hrs post-procedural, 2 velocities: carotid - femoral and carotid - radial);
* in-hospital and one month follow-up MACE.

ELIGIBILITY:
Inclusion Criteria:

* adults with ST elevation Myocardial Infarction (<12h) diagnostic confirmed;
* included in the Romanian National Programme of Primary Percutaneous Revascularisation (for who the Guidelines recommend primary PCI);

Exclusion Criteria:

* patients who do not sign informed consent for primary PCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria: study population consists of consecutive patients admitted with acute myocardial infarction (<12h) diagnostic confirmed;
  * included in the Romanian National Programme of Primary Percutaneous Revascularisation (for who the Guidelines recommend primary PCI);
  * have read and signed standard informed consent for angiography in AMI;
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hydration Status in Acute Myocardial Infarction Patients (before and after p PCI) | 2 years
  Assessment of hydration status through body composition monitoring BCM before and after coronary intervention

SECONDARY OUTCOMES:
Renal Artery Stenosis | 2 years
  Assessment of renal artery stenosis incidence in consecutive AMI patients;

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Professor, Principal Investigator — Grigore T. Popa University of Medicine and Pharmacy
Locations (1):
- Cardiovascular Diseases Institute - IASI, Iași, Iaşi, Romania